CLINICAL TRIAL: NCT01113931
Title: Safety and Efficacy of WC2031 Versus Vibramycin for the Treatment of Uncomplicated Urogenital Chlamydia Trachomatis Infection: A Randomized, Double-blind, Double-dummy, Active-controlled, Multicenter Study
Brief Title: Treatment of Chlamydia Infection Comparing WC2031 Tablets With Vibramycin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-04809
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2011-12

CONDITIONS: Urogential Chlamydia Trachomatis Infection
Keywords: Chlamydia
MeSH Terms: conditions — Chlamydia Infections | interventions — Doxycycline; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline Hyclate 200 mg tablet (Experimental): Once daily
  Interventions: Drug: Doxycyline Hyclate tablet
- Vibramycin 100 mg capsule (Active Comparator): Twice daily
  Interventions: Drug: Vibramycin (doxycyline hyclate) capsule

INTERVENTIONS:
Drug: Doxycyline Hyclate tablet — 200 mg tablet, once daily for 7 days
  Other Names: WC2031
  Arms: Doxycycline Hyclate 200 mg tablet
Drug: Vibramycin (doxycyline hyclate) capsule — 100 mg capsule, twice daily for 7 days, over-encapsulated
  Other Names: doxycycline
  Arms: Vibramycin 100 mg capsule

SUMMARY:
Evaluate the clinical efficacy and safety of WC2031 200 mg tablets taken orally once a day for 7 days versus Vibramycin (doxycycline) 100 mg capsules taken orally twice a day for 7 days, for the treatment of uncomplicated urogenital Chlamydia trachomatis infection. Primary efficacy endpoint is microbiological cure at Day 28. Safety assessments are adverse events, changes in vital signs and laboratory test results.

ELIGIBILITY:
Inclusion Criteria:

* 19-45 years of age, male or female
* presumed diagnosis of urogenital C. trachomatis infection
* use condoms during sexual activity during study (enrollment thru day 28)

Exclusion Criteria:

* Clinical diagnosis pelvic inflammatory disease or epididymitis at baseline
* Diagnosis of N. gonorrhoea
* HIV infection
* Active Hepatitis B or C infection
* Prior hysterectomy (partial or total)
* Treatment with antimicrobial therapy with known activity against urogenital C. trachomatis within 28 days of enrollment

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 495 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Caminis, MD, Study Director — Warner Chilcott
Locations (41):
- United States (41):
  - Research Site, Birmingham, Alabama
  - Research Site, Foley, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Fresno, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Boca Raton, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Margate, Florida
  - Research Site, North Miami, Florida
  - Research Site, South Miami, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Arkansas City, Kansas
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Marrero, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Fall River, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington

REFERENCES:
- [Derived] Geisler WM, Koltun WD, Abdelsayed N, Burigo J, Mena L, Taylor SN, Batteiger BE, Thurman AR, Hook EW 3rd, Vaughn TA, Annett MP, Muenzen RA, Caminis J. Safety and efficacy of WC2031 versus vibramycin for the treatment of uncomplicated urogenital Chlamydia trachomatis infection: a randomized, double-blind, double-dummy, active-controlled, multicenter trial. Clin Infect Dis. 2012 Jul;55(1):82-8. doi: 10.1093/cid/cis291. Epub 2012 Mar 19. PMID 22431798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period began 7 Apr '10
Groups:
- Doxycycline Hyclate: Morning: 1 200 mg tablet doxycycline hyclate and 1 placebo Vibramycin capsule, Evening: 1 placebo Vibramycin capsule
- Vibramycin: Morning: 1 over-encapsulated 100 mg Vibramycin tablet and 1 placebo doxycycline hyclate table, Evening: 1 over-encapsulated 100 mg Vibramycin tablet
Period: Overall Study
Arm/Group | Doxycycline Hyclate | Vibramycin
Started | 247 | 248
Safety Population | 246 (1 subject did not take any study medication) | 248
mITT Population | 188 | 190
Completed | 228 | 231
Not Completed | 19 | 17
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 12 | 9
Not completed — Various | 2 | 4
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline Hyclate | Vibramycin | Total
Number analyzed (Participants) | 247 | 248 | 495
Age Continuous [Mean (Standard Deviation); unit: years] — mITT Population
  years | 24.1 (4.9) | 23.9 (4.9) | 24.0 (4.9)
Age, Customized [Number; unit: participants] — mITT Population
  participants
    <30 years | 163 | 170 | 333
    Between 30 and 40 years | 22 | 18 | 40
    >40 years | 3 | 2 | 5
Gender [Number; unit: participants] — mITT Population
  participants
    Female | 115 | 118 | 233
    Male | 73 | 72 | 145
Ethnicity (NIH/OMB) [Number; unit: Participants] — mITT Population
  Participants
    Hispanic or Latino | 33 | 44 | 77
    Not Hispanic or Latino | 155 | 146 | 301
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: Participants] — mITT Population
  Participants
    American Indian or Alaska Native | 2 | 1 | 3
    Asian | 3 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
    Black or African American | 109 | 104 | 213
    White | 61 | 73 | 134
    More than one race | 10 | 10 | 20
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 247 | 248 | 495

OUTCOME MEASURES:

1. Primary Outcome: Microbiological Cure Rate
Description: Percentage of Subjects in mITT Population with Microbiological Cure defined as a negative result for C. trachomatis as determined by GP AC2 NAAT (Gen-Probe Aptima Combo 2 Nucleic Acid Amplification Test) at Day 28
Time Frame: Day 28
Population: mITT Population - all randomized subjects who had positive NAAT for C. trachomatis at Baseline and took at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants cured
Arm/Group | Doxycycline Hyclate | Vibramycin
Number analyzed (Participants) | 157 | 168
percentage of participants cured | 94.9 [91.5 to 98.3] | 94.6 [91.2 to 98.0]
Statistical Analysis 1: Comparison: Doxycycline Hyclate vs Vibramycin; The planned sample size of 480 randomized subjects ensured that approximately 200 subjects per group were included in the primary efficacy analyses. The 20% rate of exclusion was to account for subjects who had a negative test for urogenital C. trachomatis at the Baseline visit; Test type: Superiority or Other; Difference in Percent Cure Rates = 0.3, 95% CI 2-sided [-4.6 to 5.1]

2. Secondary Outcome: Microbiological Cure and Clinical Cure of C. Trachomatis, Day 28, Clinically Evaluable Population, Percentage Participants Cured
Description: Microbiological cure (defined as a negative result for urogenital C. trachomatis, determined by GP AC2 NAAT/Gen-Probe Aptima Combo 2 Nucleic Acid Amplification Test and clinical cure (for males defined as resolution of baseline signs/symptoms of dysuria, urethral pruritus and urethral discharge, and resolution of exam finding of urethral discharge; for females resolution of exam finding of endocervical discharge) at Day 28
Time Frame: End of Study (Day 28)
Population: Clinically Evaluable Population
Measure: Number; unit: Percentage Particpants Cured
Arm/Group | Doxycycline Hyclate | Vibramycin
Number analyzed (Participants) | 69 | 83
Percentage Particpants Cured | 80.0 | 68.6

3. Secondary Outcome: Microbiological Cure C. Trachomatis and M. Genitalium, M. Genitalium Coinfected Population, Day 28, Percentage Participants Cured
Description: Percentage Subjects Cured of both M. genitalium and C. trachomatis M. genitalium co-infected population: microbiological cure for both at Day 28, defined as negative PCR (polymerase chain reaction) for M. genitalium and negative GP AC2 NAAT (Gen-Probe Aptima Combo 2 Nucleic Acid Amplification test) for C. trachomatis at Day 28
Time Frame: End of Study (Day 28)
Population: M. genitalium Coinfected Population
Measure: Number; unit: Percentage Participants Cured
Arm/Group | Doxycycline Hyclate | Vibramycin
Number analyzed (Participants) | 15 | 12
Percentage Participants Cured | 38.5 | 18.2

4. Secondary Outcome: Microbiological Cure C. Trachomatis, N. Gonorrhoea Negative Population, Day 28, Percentage Participants Cured
Description: Percentage Participants cured in N. gonorrhoea Negative Population: cured defined as both microbiological cure (negative result for urogenital C. trachomatis, determined by GP AC2 NAAT/Gen-Probe Aptima Combo 2 Nucleic Acid Amplification test) and clinical cure (males defined as resolution of baseline signs/symptoms of dysuria, urethral pruritis and urethral discharge, and resolution of exam finding of urethral discharge; females - resolution of exam finding of endocervical discharge) at Day 28
Time Frame: Day 28
Population: N. gonorrhoea Population. Only subjects with an evaluable outcome are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage Participants Cured
Arm/Group | Doxycycline Hyclate | Vibramycin
Number analyzed (Participants) | 187 | 186
Percentage Participants Cured | 94.9 [91.4 to 98.3] | 94.6 [91.2 to 98.0]
Statistical Analysis 1: Comparison: Doxycycline Hyclate vs Vibramycin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Difference in Percent Cure Rates = 0.2, 95% CI 2-sided [-4.6 to 5.1]

ADVERSE EVENTS:
Time Frame: 28 day treatment period
Arm/Group | Doxycycline Hyclate | Vibramycin
Serious Adverse Events (participants affected / at risk) | 0/246 | 0/248
Other Adverse Events (participants affected / at risk) | 84/246 | 129/248
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline Hyclate (N=246) | Vibramycin (N=248)
Nausea (Gastrointestinal disorders) | 33 (33) | 51 (51)
Vomiting (Gastrointestinal disorders) | 20 (20) | 30 (30)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 11 (11)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (5) | 13 (13)
Vaginitis Bacterial (Infections and infestations) | 8 (8) | 5 (5)
Vulvovaginal Mycotic Infection (Infections and infestations) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less